CLINICAL TRIAL: NCT00869258
Title: Phase II Study for Inoperable Non-Metastatic Pancreatic Cancer (Stage IVA) With Neoadjuvant Gemzar, Taxotere and Xeloda (GTX), and Radiation With Gemzar
Brief Title: Study for Inoperable Non-Metastatic Pancreatic CA (Stage IVA) With Neoadjuvant GTX, and Radiation With Gemzar
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAB8630; GTX IVA (Other: protocol)
Record Dates: First submitted 2009-03-23; First posted 2009-03-25 (Estimated); Results first posted 2016-06-22 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-05

CONDITIONS: Pancreatic Cancer Stage IVA
Keywords: Pancreatic cancer; Gemcitabine; Docetaxel; Capecitabine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Docetaxel; Capecitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GTX and Radiation Therapy with Gemzar (Experimental): Chemotherapy Treatment with Gemcitabine, Docetaxel, and Capecitabine:
  A cycle of chemotherapy is made up of 21 days. During each cycle patients will take Xeloda® twice a day for 14 days followed by a rest period of 7 days. On day 4 and 11 (+/- 2 days) of each 21-day cycle patients will also receive Gemzar and Taxotere.
  Weekly Radiation Therapy with Low-Dose Gemzar Chemotherapy:
  After completing a total of 3 cycles of GTX chemotherapy each patient will receive 5 weeks of standard radiation therapy in combination with low-dose Gemzar chemotherapy.
  Interventions: Drug: Gemcitabine, docetaxel, and capecitabine; Radiation: Radiation therapy with gemzar

INTERVENTIONS:
Drug: Gemcitabine, docetaxel, and capecitabine — Day 1-14: Capecitabine 1500 mg/m2/day (+/- 2days) Day 4 and 11: Gemcitabine 750 mg/m2/day (+/- 2days) Day 4 and 11: Docetaxel 30 mg/m2/day (+/- 2 days) Two week treatment regimen is followed by one week off, repeated for a total of 3 cycles
  Other Names: Gemzar; Taxotere; Xeloda; GTX
Radiation: Radiation therapy with gemzar — Starting on week 12 +/- 5 days radiation therapy will be given in the standard manner over 5 weeks with daily radiation fractions Monday through Friday. Once a week gemcitabine will be given IV over 30 minutes at 250-300 mg/m2
  Other Names: Radiation therapy with gemcitabine

SUMMARY:
The purpose of this study is to determine whether an experimental drug combination consisting of Gemzar®, Taxotere®, and Xeloda®, (called GTX) when followed by radiation therapy plus low-dose Gemzar, is safe and effective in treating advanced pancreatic cancer and to study and enhance the utility of PET scans in the evaluation of patients with pancreatic cancer.

DETAILED DESCRIPTION:
The evolution of our regimen, consisting of Gemzar, Taxotere and Xeloda (oral 5FU) (GTX), was carefully developed over the past three years from laboratory and clinical work. Initially, in collaboration with Dr. William Sherman of the Division of Medical Oncology we assessed the clinical effects of two agents, Gemzar and Taxotere in pancreatic cancer patients. In our in vitro studies we found that as single agents these drugs (Gemzar and Taxotere) were minimally effective against pancreatic carcinoma lines, which expressed mutant p53 and activated mutated ras. Activated or mutant ras is found in approximately 95% of all pancreatic carcinomas. However, when the agents were added together in tissue culture experiments we found that their activity was additive. The clinical study performed at Columbia Presbyterian Medical Center demonstrated a 27% objective response rate by CT scan including one complete response with intent to treat analysis of all 15 patients within the study. The majority of these patients had metastatic liver disease and a minority had inoperable pancreatic carcinoma without liver metastases. Though this was a small single arm, single institution study it did suggest a trend towards improved responses in patients with this disease when these two agents were combined. In addition, valuable lessons were learned from the in vitro work with Gemzar and Taxotere. Importantly, we found that this combination was equally toxic to mutant and wild type p53 pancreatic cancer cells, as well as to cells with mutant ras. Also, docetaxel pharmacokinetics are more favorable and have distinct advantages over the use of the other taxane known as paclitaxel. They are the following: 1) Taxotere enters tumor cells more efficiently than paclitaxel because it is more lipophilic; 2) Taxotere is not pumped out by the cell by P-glycoprotein as efficiently as paclitaxel; 3) Taxotere' half life was significantly longer than that of paclitaxel such that a 60 minute infusion of Taxotere gives you approximate pharmacokinetics as paclitaxel when administered as a 24 hour continuous infusion. These laboratory studies from the literature formed the rationale for our use of Taxotere (docetaxel) instead of paclitaxel.

After our initial clinical and laboratory study we went back to the laboratory to investigate further some of the properties of Gemcitabine, Taxotere added to Xeloda (5-DFUR) in vitro to maximize biochemical synergy and to minimize toxicity. We found important characteristics of these drug combinations against pancreatic cancer cells that have been synthesized into the current protocol. We found that there was sequence specificity for these drugs in that 5-DFUR should precede Gemzar by 72 to 96 hours and Gemzar should be added before Taxotere to achieve maximum synergy. Taxotere cytotoxicity was dose dependent up to 20 nM but then no further cell kill was obtained past that point. This would mean that one would not need to use high dose Taxotere in a regimen because it would be doubtful whether increased doses would obtain further cell kill in a linear scale.

We investigated many different combinations of these 3 agents in the laboratory to determine the best combination to achieve biochemical synergy while decreasing the concentration of each drug and not lose anti-tumor effect so as to decrease toxicity to patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of pancreas localized to the pancreas, small bowel, stomach and/or encasing the superior mesenteric artery, vein or portal vein. (a.k.a. Stage IV A).
* No prior chemotherapy for their pancreatic cancer or radiation to the area of the tumor.
* Measurable disease: Any mass reproducibly measurable in two perpendicular diameters by x-ray, physical examination, CT or MRI scans.
* Ineligible for other high priority national or institutional studies
* Whipple surgery not allowed. Prior surgery is allowed as long as it was not pancreatic resection (i.e. Whipple surgery) and the time from surgical recovery is greater than three weeks.
* Non pregnant females who are not breast feeding with a negative serum β-HCG test within 1 week of starting the study. Men and women of childbearing potential must be willing to consent to using effective contraception while on treatment and for a reasonable period thereafter.
* Clinical Parameters

  * Life expectancy > 2 months.
  * Age 18 to 70 years old
  * Performance status 0-2 (ECOG). (See Appendix IV)
  * Peripheral Neuropathy must be < grade 1
  * Able to tolerate oral medications
  * Absolute Neutrophil Count > 1,500 μl
  * White Blood Count > 3,000/μl
  * Platelet count > 100,000/μl
  * BUN < 1.5 x normal
  * Creatinine < 1.5 normal
  * Hemoglobin > 8.0 g/dl
  * Serum Albumin > 2.5 mg/dl
  * Total Bilirubin < 5.0 mg/dl
  * SGOT, SGPT, Alkaline Phosphatase < 4.0 x ULN

Exclusion Criteria:

* Hypersensitivity: Patients with a history of severe hypersensitivity reaction to Taxotere® or other drugs formulated with polysorbate 80 must be excluded.
* Informed Consent: Each patient must be completely aware of the nature of his/her disease process and must willingly give consent after being informed of the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts.
* Prior malignancies in last 5 years other than: curatively treated carcinoma in-situ of the cervix, non-melanoma skin cancer, prostate or DCIS (ductal carcinoma in-situ) previously treated successfully (cancer free)
* No serious medical or psychiatric illness preventing informed consent or intensive treatment (e.g., serious infection).
* Patients known to have HIV will be excluded.
* Patients cannot have received any prior investigational agent/therapy, nor will they be allowed any investigational agent/therapy while on protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Fine, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Unknown.

REFERENCES:
- [Derived] Sherman WH, Hecht E, Leung D, Chu K. Predictors of Response and Survival in Locally Advanced Adenocarcinoma of the Pancreas Following Neoadjuvant GTX with or Without Radiation Therapy. Oncologist. 2018 Jan;23(1):4-e10. doi: 10.1634/theoncologist.2017-0208. Epub 2017 Dec 6. PMID 29212734

RESULTS

PARTICIPANT FLOW:
Groups:
- GTX and Radiation Therapy With Gemzar: Chemotherapy Treatment with Gemcitabine, Docetaxel, and Capecitabine (GTX) and weekly radiation therapy with low-dose Gemzar chemotherapy.
Period: Overall Study
Arm/Group | GTX and Radiation Therapy With Gemzar
Started | 32
Completed | 31
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | GTX and Radiation Therapy With Gemzar
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 22
  More than one race | 5
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Conversion Rate of Inoperable to Operable
Description: Data was not analyzed because original PI left institution before data analysis was completed.
Time Frame: 10 weeks
Arm/Group | GTX and Radiation Therapy With Gemzar
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | GTX and Radiation Therapy With Gemzar
Serious Adverse Events (participants affected / at risk) | 4/32
Other Adverse Events (participants affected / at risk) | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTX and Radiation Therapy With Gemzar (N=32)
Fever (Infections and infestations) | 1 (1)
Clogged Common Bile Duct (CBD) Stent (Hepatobiliary disorders) | 1 (1)
Gastrointestinal (GI) Bleed (Gastrointestinal disorders) | 1 (1)
Irritable Bowel (Gastrointestinal disorders) | 1 (1)
Gallbladder Issues and Fever (Gastrointestinal disorders) | 1 (1)
Stent Replacement and Possible Biliary Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GTX and Radiation Therapy With Gemzar (N=32)
Fatigue (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Infectious Colitis (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Abnormal Creatinine Level (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (General disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Metabolism and nutrition disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes